CLINICAL TRIAL: NCT01874392
Title: Feasibility Study Using Zone-MPC Controller (Zone-Model Predictive Control) and Health Monitoring System (HMS) and Technosphere® Insulin Inhalation System From MannnKind Corp.
Brief Title: Feasibility Study Using Zone-MPC Controller, HMS and Technosphere® Insulin Inhalation System From MannnKind Corp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JDRF 17-2010-765
Record Dates: First submitted 2013-05-14; First posted 2013-06-11 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T1DM (Experimental): Adults aged 21-65 years with type 1 diabetes mellitus for at least one year who are using an insulin infusion pump with rapid-acting insulin for at least six months
  Interventions: Drug: Investigational inhaled insulin (Technosphere); Device: Artificial Pancreas (AP) device (APS©)

INTERVENTIONS:
Drug: Investigational inhaled insulin (Technosphere) — by MannKind Corp. IND 61,729
  Other Names: Technosphere® Insulin Inhalation System (Gen2C inhaler)
Device: Artificial Pancreas (AP) device (APS©) — Device includes:
  * OneTouch® Ping® Glucose Management System with modified Meter-Remote from Animas® Corp or the OmniPod® Insulin Management System from Insulet Corp.
  * Dexcom® G4® CGM System (CGM) from Dexcom® Corp
  * Control algorithm: zone-Model Predictive Control (zone-MPC) with safety Health Monitoring System (HMS)
  Other Names: Artificial Pancreas System platform (APS©) from the University of California, Santa Barbara and SDRI

SUMMARY:
This clinical trial is a feasibility study to assess the performance of an Artificial Pancreas (AP) device using the Artificial Pancreas System (APS©) platform for subjects with type 1 diabetes using rapid-acting insulin as well as preprandial inhaled insulin (Technosphere® Insulin Inhalation System by MannKind Corporation). The goal of this proposed study is to explore the feasibility of using multiple insulin delivery routes in order to mimic the physiology of both first- and second-phase insulin secretion. The intent is to exploit the rapid action achieved by inhaled insulin to compensate for part of the meals and utilize the conventional subcutaneous route for management of basal insulin and as second-phase meal-related insulin.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least one year and using an insulin pump for at least 6 months with commercially available rapid actin insulin
* The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
* Age 21 to 65 years
* For females, not currently known to be pregnant or nursing
* HbA1c between 5.0% and 10%, as measured with DCA2000 or equivalent device
* Forced expiratory volume in 1 second (FEV1) ≥ 70% Third National Health and Nutrition Examination Survey (NHANES III) predicted
* Forced vital capacity (FVC) ≥70% NHANES III predicted
* Forced expiratory volume in 1 second as a percentage of forced vital capacity(FEVl/FVC)≥NHANES III lower limit of normal (LLN)
* Willing to perform the calibration of the study CGMs using a finger stick only and willing to follow instructions for insulin pump and CGM wear.
* Willing to use the study CGM and study insulin pump during closed-loop.
* Able to and agrees to avoid the following medication starting 24 hours before sensor wear through completion of CRC visit: acetaminophen, and pseudoephedrine.
* An understanding of and willingness to follow the protocol and sign the informed consent.

Exclusion Criteria:

* Pregnancy (as determined by a positive blood pregnancy test performed in females of childbearing capacity during screening visit and urine test at time of admission for in-patient visit) or nursing mother.
* Diabetic ketoacidosis in the past 6 months prior to enrollment requiring emergency room visit or hospitalization
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
* Current treatment for a seizure disorder;

  o Subjects with a history of seizures may be included in the study if they receive written clearance from their neurologist
* Cystic fibrosis
* Active infection
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as cognitive deficit.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation, including subjects not able to read or write.
* Coronary artery disease or heart failure. oSubjects with a history of coronary artery disease may be included in the study if they receive written clearance from their cardiologist
* Presence of a known adrenal disorder
* Active coronary artery disease or heart failure
* Active gastroparesis
* If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
* Uncontrolled thyroid disease

  o Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment
* Abuse of alcohol
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the exercise protocol
* Current use of a beta blocker medication
* Laboratory results:

  * Hematocrit < 30% or >55%
  * A1C > 10%
  * Abnormal liver or renal function (Transaminase >2 times the upper limit of normal, Creatinine> 1.5 mg/dL)
  * Labs drawn at screening visit or within one month prior to screening (for other purposes) will suffice for enrollment purposes related to hematocrit
* Subject has skin conditions that, in the determination of the investigator, would preclude wearing the study devices (infusion set and sensor), in the abdomen. Examples include but are not limited to: psoriasis, burns, scaring, eczema, tattoos, and significant hypertrophy at sites of device wear; any known allergy to medical adhesives.
* Currently on long-term treatment using prednisone.
* If subject had been on short term treatment of prednisone, defer enrollment until underlying condition and prednisone treatment have resolved.
* Allergy to study drug, food or other study material
* History of asthma, COPD (chronic obstructive pulmonary disease), or any other clinically relevant chronic lung disease
* Respiratory track infection within 4 weeks before screening
* Clinically significant screening ECG, physical examination, laboratory test, or vital sign abnormality
* Exposure to any investigational drug within 30 days.
* History of malignancy within the 5 years before screening (other than basal cell carcinoma)
* Inability, in the opinion of the investigator, to adequately inhale Technosphere® Inhalation powder
* Abnormal spirometry
* Currently smoking or discontinued smoking (including cigarettes, cigars, pipes) over the past 6 months.
* Highly sensitive to insulin: insulin-to-carbohydrate ratio I:C > 1:12.
* Current participation in another investigational trial (unless participation to original protocol of IDE G110093) or has previously participated to this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Zisser, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

REFERENCES:
- [Result] Zisser H, Dassau E, Lee JJ, Harvey RA, Bevier W, Doyle FJ 3rd. Clinical results of an automated artificial pancreas using technosphere inhaled insulin to mimic first-phase insulin secretion. J Diabetes Sci Technol. 2015 May;9(3):564-72. doi: 10.1177/1932296815582061. Epub 2015 Apr 21. PMID 25901023

RESULTS

PARTICIPANT FLOW:
Groups:
- T1DM: Adults aged 21-65 years with type 1 diabetes mellitus for at least one year who are using an insulin infusion pump with rapid-acting insulin for at least six months
  Investigational inhaled insulin (Technosphere): by MannKind Corp. IND 61,729
  Artificial Pancreas (AP) device (APS©): Device includes:
  * OneTouch® Ping® Glucose Management System with modified Meter-Remote from Animas® Corp or the OmniPod® Insulin Management System from Insulet Corp.
  * Dexcom® G4® CGM System (CGM) from Dexcom® Corp
  * Control algorithm: zone-Model Predictive Control (zone-MPC) with safety Health Monitoring System (HMS)
Period: Overall Study
Arm/Group | T1DM
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | T1DM
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Test the Safety of the AP Device While the Subject is Under Close Medical Supervision in the Clinical Research Center (CRC) Setting.
Description: This objective will be assessed by subjecting the AP device (combined with the Technosphere® Insulin Inhalation Powder) and the subject to several challenging situations, such as meals, exercise, and nocturnal period. The study will evaluate the percent of time the glucose level of the subject remains within Target range 5 hours after meal: [70-180] mg/dL.
Time Frame: 5 hours
Measure: Median (Inter-Quartile Range); unit: percentage time in range (70 - 180 mg/dL
Arm/Group | T1DM
Number analyzed (Participants) | 9
percentage time in range (70 - 180 mg/dL | 81.6 [72.5 to 85.0]

2. Primary Outcome: Test the Safety of the AP Device While the Subject is Under Close Medical Supervision in the Clinical Research Center (CRC) Setting.
Description: This objective will be assessed by subjecting the AP device (combined with the Technosphere® Insulin Inhalation Powder) and the subject to several challenging situations, such as meals, exercise, and nocturnal period. The study will evaluate the percent of time the glucose level of the subject remains within Target range for the entire study: [80-140] mg/dL
Time Frame: 25-28 hours
Measure: Median (Inter-Quartile Range); unit: percentage time in range(80-140mg/dL)
Arm/Group | T1DM
Number analyzed (Participants) | 9
percentage time in range(80-140mg/dL) | 67.5 [48.5 to 73.1]

3. Primary Outcome: Test the Safety of the AP Device While the Subject is Under Close Medical Supervision in the Clinical Research Center (CRC) Setting
Description: This objective will be assessed by subjecting the AP device (combined with the Technosphere® Insulin Inhalation Powder) and the subject to several challenging situations, such as meals, exercise, and nocturnal period. The study will evaluate the percent of time the glucose level of the subject remains within Target range during exercise: [70-150] mg/dL
Time Frame: 30 minutes
Measure: Median (Inter-Quartile Range); unit: percentage time in range (70-150 mg/dL)
Arm/Group | T1DM
Number analyzed (Participants) | 9
percentage time in range (70-150 mg/dL) | 94.4 [91.6 to 94.4]

4. Primary Outcome: Test the Safety of the AP Device While the Subject is Under Close Medical Supervision in the Clinical Research Center (CRC) Setting
Description: This objective will be assessed by subjecting the AP device (combined with the Technosphere® Insulin Inhalation Powder) and the subject to several challenging situations, such as meals, exercise, and nocturnal period. The study will evaluate the percent of time the glucose level of the subject remains within Target range 3 hours after exercise: [70-150] mg/dL
Time Frame: 3 hours
Measure: Median (Inter-Quartile Range); unit: percentage time in range (70-150 mg/dL)
Arm/Group | T1DM
Number analyzed (Participants) | 9
percentage time in range (70-150 mg/dL) | 94.4 [91.6 to 94.4]

5. Primary Outcome: Test the Safety of the AP Device While the Subject is Under Close Medical Supervision in the Clinical Research Center (CRC) Setting.
Description: This objective will be assessed by subjecting the AP device (combined with the Technosphere® Insulin Inhalation Powder) and the subject to several challenging situations, such as meals, exercise, and nocturnal period. The study will evaluate the percent of time the glucose level of the subject remains within Overnight target range: [70-180] mg/dL
Time Frame: 7 hours overnight
Measure: Median (Inter-Quartile Range); unit: percentage time in range (70 - 180 mg/dL
Arm/Group | T1DM
Number analyzed (Participants) | 9
percentage time in range (70 - 180 mg/dL | 100 [95.2 to 100]

6. Secondary Outcome: Test the Benefits of the AP Device Combined With the Technosphere® Insulin Powder System
Description: To evaluate the performance of the AP device combined with the Technosphere® Insulin Powder System after dinner by measuring the postprandial excursion of blood glucose.
Time Frame: 150 minutes
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | T1DM
Number analyzed (Participants) | 9
mg/dL | 64 [30 to 120]

7. Secondary Outcome: Test the Benefits of the AP Device Combined With the Technosphere® Insulin Powder System
Description: To evaluate the performance of the AP device combined with the Technosphere® Insulin Powder System after breakfast by measuring the postprandial excursion of blood glucose
Time Frame: 120 minutes
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | T1DM
Number analyzed (Participants) | 9
mg/dL | 61 [56 to 85]

ADVERSE EVENTS:
Time Frame: 25-28 hours
Arm/Group | T1DM
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT01874392/Prot_SAP_000.pdf